CLINICAL TRIAL: NCT05376761
Title: Median Effective Concentration (EC50) of Dexmedetomidine in Deep Brain Stimulation Implantation of Patients With Parkinson's Disease
Brief Title: EC50 of Dexmedetomidine in Deep Brain Stimulation Implantation of Patients With Parkinson's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Director of Anesthesiology Department, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: xsn20220314
Record Dates: First submitted 2022-05-08; First posted 2022-05-17 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: PD - Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DEX for STN-DBS (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — The loading dose of DEX (0.5 µg/kg) is transfused intravenously within 15min.The maintaining concentration of DEX, which is started at 0.3 µg/kg/h in the first patient, is determined by the NRMS in the MER signal of the previous patient according to the up and down sequence. If the NRMS is higher than 2.0, a positive response is defined and the concentration of DEX will be added by 0.05µg/kg/h in the next patient. A negative response is defined as NRMS lower than 2.0, and in such cases the concentration of DEX is reduced by 0.3 µg/kg/h.

SUMMARY:
Dexmedetomidine (DEX) sedation is widely used in deep brain stimulation implantation (DBSI) of patients With Parkinson's disease. However, intraoperative application of DEX may affect the discharge activity of deep brain nuclei and reduce the discharge frequency of Subthalamic nucleus (STN) neurons. At present, there is still a lack of prospective intervention research to explore the optimal dose that does not affect MER mapping in patients with Parkinson's disease. The present study uses the Dixon and Massey up-and-down method to analyze the EC50 of DEX in patients with PD undergoing STN-DBS sedation, to clarify the balance meets the sufficient comfort of patients without affecting the accurate target of MER and the optimal dosage of DEX for boundary recognition.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is an effective treatment to improve the motor symptoms of Parkinson's disease (PD). Subthalamic nucleus (STN) is one of the most commonly used targets in the treatment of PD-DBS. The accuracy of the final implantation position of deep brain electrodes is the key to the success of surgery.

Sedation-Awake-Sedation anesthesia is widely used in DBS. Dexmedetomidine (DEX) mainly acts on the central locus coeruleus nucleus and spinal cord α receptor, which has sedative and analgesic effect and little respiratory inhibition. DEX can produce natural non eye movement sleep that is conducive to the recovery of the body. Within a certain dose range, patients are easy to wake up and have the characteristics of conscious sedation. Patients can make corresponding actions according to the instructions of neurosurgeons and cooperate with doctors to complete the operation. Its sedative safety has been confirmed.

However, intraoperative application of DEX may delay the recovery of cognitive function, affect the discharge activity of deep brain nuclei and reduce the discharge frequency of STN neurons, even after stopping the use of sedatives. The result may be related to the residual effect of sedatives. DEX can reduce the activity of STN neurons in a dose-dependent manner. A smaller dose of DEX may not meet the effects of surgical sedation and analgesia, and the effect of high concentration is better than that of low concentration. Some existing studies have recommended a reasonable dose range of DEX for DBS, but these studies have a small number of research populations, and of great heterogeneity in target selection, anesthetic dose and strategy. At present, there is still a lack of prospective intervention research to explore the optimal dose that the application of DEX sedation does not affect MER mapping in patients with Parkinson's disease. The present study uses the up and down method to analyze the EC50 and EC95 of DEX in patients with PD undergoing STN-DBS sedation, to clarify the balance meets the sufficient comfort of patients without affecting the accurate target of MER and the optimal dosage of DEX for boundary recognition.

ELIGIBILITY:
Inclusion Criteria:

1. 50-80 years old, ASA grade II-III;
2. Bilateral STN-DBS of patients with Parkinson's disease;
3. Signed informed consent.

Exclusion Criteria:

1. Obstructive sleep apnea;
2. BMI > 30kg/m2;
3. Estimated difficult airway;
4. Severe preoperative anxiety;
5. Serious dysfunction of important organs such as heart, liver and kidney;
6. previous allergy to dexmedetomidine;
7. Pregnant or lactating women.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
EC50 and the corresponding 95%CI of DEX applied to PD patients undergoing STN-DBS are determined by the up and down method according to the normalized root mean square(NRMS) value of the MER sampled signal. | during MER recording
  We use the root mean square (RMS) value of the MER sampled signal recorded by the electrode, measured in volts, as the main parameter for evaluating electrode position. RMS values change with the electrode properties and other external drives related to the operating room; therefore, it is crucial to normalize the RMS to comparable values. Thus, each session's RMS in a trajectory is divided by the mean RMS of the first five stable sessions in the same trajectory. This normalized RMS (NRMS) is found to be a good measure as it reflects the relative change in the total power of the signal, which elevates dramatically entering the STN.
  If the NRMS is higher than 2.0, a positive response is defined and the concentration of DEX will be added by 0.05µg/kg/h in the next patient. A negative response is defined as NRMS lower than 2.0, and in such cases the concentration of DEX is reduced by 0.3 µg/kg/h.

SECONDARY OUTCOMES:
STN pass length (mm) | during MER recording
  For STN identification and length, recordings within the thalamus, zona incerta, STN, and SNr are identified by an experienced neurophysiologist intraoperatively and reclassified independently offline. The STN pass length is determined as the distance from entry to exit of the STN based on the significant, clear increase in baseline unit activity and FR changes unique to STN.

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, MD, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan hospital, Beijing, Beijing Municipality, China